CLINICAL TRIAL: NCT06370000
Title: REMAIN1: Relapse Prevention With Maintenance Oral Azacitidine in Transplant Eligible Patients With Acute Myeloid Leukemia Not Proceeding to Transplant Due to Racial or Socioeconomic Disparities
Brief Title: Oral Azacitidine in Transplant-Eligible Patients With Acute Myeloid Leukemia (AML) Suffering From Health-Inequality
Acronym: REMAIN1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23-20817; HM20029540 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Azacitidine (Experimental): Starting dose is oral azacitidine 300 mg orally once daily with or without food days 1-14 in a 28-day cycle
  Interventions: Drug: Oral Azacitidine

INTERVENTIONS:
Drug: Oral Azacitidine — Oral Azacitidine, 300mg PO Daily during days 1-14 of a 28 day cycle for up to 6 cycles.

SUMMARY:
Test feasibility of an oral maintenance strategy for transplant eligible AML patients in first CR who are medically underserved or have a disadvantage in the CDC SDOH domains

DETAILED DESCRIPTION:
This is a non-randomized open-label single institution pilot study that will evaluate the feasibility, toxicity, and efficacy of maintenance oral azacitidine in medically transplant eligible non-FMS-like tyrosine kinase 3 (FLT3) mutated AML patients with a disadvantage in at least 1 of the 5 key Center for Disease Control and Prevention (CDC) defined social determinants of health (SDOH) domains that are preclusive to transplant at time of study enrollment, as identified either by the patient or a member of the healthcare team.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-Acute Promyelocytic (APL) FLT3 negative AML and have completed induction and consolidation as defined by the treating physician and must be in complete response (CR), Complete response with partial hematologic recovery (CRh), or Complete response with incomplete count recovery (CRi) at time of study enrollment
* For patients in CR1, AML disease phenotype must be one that is considered for allo HCT in CR1 (intermediate or high risk by European Leukemia Net (ELN), MRD+ CR, slow clearance of MRD) or any AML phenotype (aside from FLT3+ and APL) in CR2 and beyond
* Medically eligible for allogeneic hematopoietic cell transplant (allo HCT) as defined by either: treating physician discretion, transplant physician discretion, or hematopoietic cell transplantation-specific Comorbidity index (HCT-CI) index of 5 or less
* Age ≥ 18 years
* Enrollment must occur within 4 months of completion of therapy
* A patient or staff identified health disparity in 1 of the 5 Centers for Disease Control (CDC) defined social determinants of health (SDOH). This may include financial difficulties, lack of caregiver support, difficulties with medical literacy, rurality, appropriate access to health care, lack of an appropriate allogeneic hematopoietic cell transplant (allo HCT) donor, substance abuse
* Patient must have adequate organ function defined as: Creatinine clearance (by Cockroft-Gault formula) greater than or equal to 29 mL/min, total bilirubin and aspartate aminotransferase/ alanine transaminase (AST/ALT) ≤ to institutional 2x upper limit of normal (except Gilbert's syndrome, which may enroll if < 2x patient's baseline total bilirubin)
* Eastern Cooperative Oncology Group (ECOG) 0,1,2,3
* Ability to take oral medications
* No history of malabsorption syndrome which, in the investigator's opinion, may inhibit absorption of oral medications
* Women of childbearing potential must consent to effective contraception during study treatment and at least 6 months following the last dose. Women who are breastfeeding are also excluded
* Male patients must consent to effective contraception during study and at least 3 months after last dose
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria A patient who meets any of the following exclusion criteria is ineligible to participate in the study.

* FMS-like tyrosine kinase 3 (FLT3 ITD) or tyrosine kinase domain (TKD) mutation
* Uncontrolled central nervous system (CNS) involvement
* History of hypersensitivity or allergic reaction to azacitidine or its components
* Stem cell transplant within previous 3 months prior to initiation of study therapy
* Uncontrolled intercurrent illness or infection
* History of prior therapy with oral azacitidine
* Female patients who are pregnant or intend to donate eggs during the study or for 6 months after receiving their last dose of study drug
* Male patients who intend to donate sperm during the course of this study or for 3 months after last dose
* Other malignancy for which the patient is currently receiving therapy (except excisable skin cancer)
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the participant's risk or limit the participant's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of completion of at least 4 cycles an oral maintenance strategy for transplant eligible AML patients in CR who are medically underserved or have a disadvantage in the CDC SDOH domains | 4 months
  The number of participants that complete at least four cycles of protocol therapy

SECONDARY OUTCOMES:
Overall survival (OS) | 3 months, and up to 2 years
  Number of participants alive at relapse, completion of treatment or removal from study.
Leukemia Free Survival (LFS) 3 months after beginning of treatment and at relapse, completion of treatment or removal from study | 3 months, and up to 2 years
  Number of participants still in remission 3 months after beginning of treatment and at relapse, completion of treatment or removal from study
Measure rates of measurable residual disease (MRD) negativity | 3 months, and up to 2 years
  The number of participants that have negative measurable residual disease (MRD) at 3 months after beginning of treatment, and completion of treatment. MRD will be measured by flow cytometry and by pathologic complete response (PCR) based molecular assay if/when target gene is available on diagnostic specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Keri Maher, DO, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data. Datasets are available on reasonable request to the author.